CLINICAL TRIAL: NCT06696352
Title: Partners for Pain & Wellbeing: A Randomized Trial of Community Supported Complementary and Integrative Health Self Management for Back Pain
Brief Title: Partners4Pain & Wellbeing: A Randomized Trial of Community Supported Complementary and Integrative Health Self-management for Back Pain
Acronym: P4P
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R33AT012309 (NIH); R33AT012309 (NIH); STUDY00017917 (Other: University of Minnesota Institutional Review Board)
Record Dates: First submitted 2024-11-05; First posted 2024-11-20 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Chronic Pain; Back Pain; Neck Pain; Self-management; Complementary Therapies
Keywords: Self-Management; Chronic Pain; Neck Pain; Low Back Pain; Complementary Therapies; Back Pain
MeSH Terms: conditions — Chronic Pain; Back Pain; Neck Pain; Low Back Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Partners4Pain (Experimental): Community-based program that focuses on evidence based mind-body tools (mindfulness, cognitive behavioral approaches) for pain self-management in addition to pain education and physical exercises.
  Interventions: Behavioral: Partners4Pain
- Keys to Wellbeing (Active Comparator): Community-based program that focuses on general health and well-being education for pain self-management in addition to pain education and physical exercises.
  Interventions: Behavioral: Keys to Wellbeing

INTERVENTIONS:
Behavioral: Partners4Pain — This is a group program that will teach participants about different things they can do to manage their pain. They will watch educational videos and do workbook activities. They will learn and practice different exercises and mind-body strategies for pain including back and neck exercises (like strengthening and stretching), mind-body exercises (like meditation, relaxed breathing, guided imagery, and muscle relaxation), problem solving, and how to communicate with others about your pain. They will also have an opportunity to take part in discussions with other group members. The program will be delivered via weekly 90 minute sessions over 9 weeks and will be offered in-person or via videoconference.
  Arms: Partners4Pain
Behavioral: Keys to Wellbeing — This is a group program that will teach participants about different things they can do to improve their health and wellbeing. Participants will watch educational videos and do workbook activities. They will learn different back and neck exercises (like strengthening and stretching) and be introduced to different health-related topics including information and tips about health, pain and wellbeing; keeping active and well; the importance of rest and relaxation; and working with meaning and purpose in your life. They will also have an opportunity to take part in discussions with other group members. The program will be delivered in weekly 90 minute sessions over 9 weeks and will be offered in-person or via videoconference.
  Arms: Keys to Wellbeing

SUMMARY:
The goal of this clinical trial is to learn how well two community-based self-management programs work in people with chronic back or neck pain. The main question it aims to answer is:

How well does a community-based self-management program teaching mind-body skills such as mindfulness and cognitive behavioral approaches (Partners4Pain) work for reducing pain intensity and interference with general activities and enjoyment of life compared to a community-based self-management program focused on general health and wellbeing (Keys to Wellbeing)?

Participants will be asked to do the following:

* Attend 2 screening visits to learn about the study and see if they meet the requirements to participate.
* Be randomly assigned to one of the two community-based self-management programs.
* Attend 9 weekly self-management program sessions (90 minutes each)
* Complete surveys about their pain and overall health at 2 months (after the programs end), 4 months, and 6 months.

Funding for the project is provided through the National Center for Complementary and Integrative Health (NCCIH) and the National Institute of Neurological Disorders and Stroke (NINDS) through the NIH HEAL Initiative (https://heal.nih.gov/), R33AT012309.

DETAILED DESCRIPTION:
This project is a full-scale, multi-level randomized hybrid effectiveness implementation trial (n=376) of 'Partners4Pain', a community supported self-management program for individuals with back or neck pain. Partners4Pain will be compared to an active control, Keys to Wellbeing. Both programs were optimized and feasibility tested in an earlier R61 pilot study of 51 individuals (NCT05786508).

Aims for the hybrid effectiveness implementation trial are:

AIM 1. To assess the relative effectiveness of Partners4Pain versus Keys to Wellbeing in terms of:

* Primary effectiveness outcomes of pain intensity and interference over 6 months using bi-monthly assessments.
* Secondary effectiveness outcomes of pain impact, self-efficacy and other HEAL outcomes.

AIM 2. To assess the impact of health factors on the effectiveness of Partners4Pain for primary and secondary outcomes through subgroup analyses which account for potential complexities between factors.

AIM 3. To describe important implementation related measures that can impact and inform sustained translation of the program with community partner organizations.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Self-reported chronic back pain (defined as pain in the low or mid back, or neck pain) which has lasted for 3 months or longer
* Score of 3 or higher on the self-reported Pain, Enjoyment of Life and General Activity scale (PEG scale - 0-10)
* Member of one or more of the following populations: American Indian/Alaska Native; Asian; Black/African American; Hispanic/Latino; Native Hawaiian/Pacific Islanders; Socioeconomically disadvantaged (annual household income less than $50,000)
* Reside within the Minneapolis/St. Paul metro region

Exclusion Criteria:

* Severe unmanaged mental illness
* Self-reported cancer with active treatment involving radiation or chemotherapy.
* Dementia - Mini Mental State Exam score of 23 or lower for those with suspicion of cognitive impairment
* Self-reported pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Pain, Interference with Enjoyment of Life and General Activity | Baseline, 2, 4, 6 months
  Measured using the Pain, Enjoyment of Life and General Activity (PEG) scale that measures average pain intensity, interference with enjoyment of life, and interference with general activity in the past week. Each item is measured on a 0 (no pain/does not interfere) to 10 numeric rating scale (pain as bad as you can imagine/completely interferes).

SECONDARY OUTCOMES:
Graded Chronic Pain Scale | Baseline, 2, 6 months
  Measured using the Graded Chronic Pain Scale-Revised (GCPS-R), a six item scale developed to differentiate mild, bothersome, and high-impact chronic pain. Two questions to identify chronic pain and high impact chronic pain; frequency of pain during the prior 3 months and frequency of limitation in activities in the prior 3 months.
Self-efficacy for Managing Chronic Conditions | Baseline, 2, 4, 6 months
  Measured using the PROMIS 4-item short forms for 1) managing daily activities; 2) managing symptoms; 3) managing emotions; and 4) managing social interactions. All Items are scored on a 5-point Likert scale (1=I am not confident at all to 5=I am very confident).
Domain Specific Life Satisfaction | Baseline, 2, 4, 6 months
  Domain-Specific Life Satisfaction is a 13-item PROMIS measure of satisfaction with various aspects of life (e.g. education, housing, family life, health, neighborhood). Agreement with statements of satisfaction for each domain are measured on a 5-point scale ranging from Not at all to Very much.
Quality of Life and Health Satisfaction | Baseline, 2, 4, 6 months
  Measured using the World Health Organizations 2-item measure which measures quality of life and satisfaction with health on a 1 to 5 scale.
Physical Functioning | Baseline, 2, 4, 6 months
  The PROMIS Physical functioning 6-item short form v2.0 which measures difficulty doing household activities and agreement with statements on health limitations in physical activities on a 1 to 5 scale.
Pain Catastrophizing | Baseline, 2, 4, 6 months
  Assessed using the Pain Catastrophizing Scale (PCS), a 6-item self-reported measure to indicate the degree to which a person may ruminate, magnify, and feel helpless about their pain. The PCS-6 measures a person's thoughts and feelings when they are experiencing pain using the 0 (not at all) to 4 (all the time) scale.
Interoceptive Awareness | Baseline, 2, 4, 6 months
  Measured using the Multidimensional Assessment of Interoceptive Awareness (MAIA) survey instrument (V2) using the 1) noticing; 2) attention regulation; 3) emotional awareness; and 4) self-regulation subscales.
Overall Improvement | Months 2, 4, 6
  Overall improvement will be assessed with the Patient Global Impression of Change (PGIC) which has participants rate their overall change from very much worse to very much improved on a 7-point scale.
Intervention Satisfaction | Months 2, 4, 6
  Assessed using a question that has participants rate their overall satisfaction ranging from completely satisfied to completely dissatisfied on a 7-point scale.
Social Isolation | Baseline, 2, 4, 6 months
  Measured using the PROMIS 4-item short form v2.0 which measures frequency of different feelings of social isolation on a 1 (Never) to 5 (Always) scale.
Healthcare Use | Baseline, 2, 4, 6 months
  Participant self report of provider visits, emergency department visits, diagnostic imaging scans, hospitalizations, injections and surgical procedures for neck and back pain.
Medication Use | Baseline, 2, 4, 6 months
  Participant self-report of over the counter and prescription medication use for back or neck pain.
Complementary Integrative Health Self-Management Use | Baseline, 2, 4, 6 months
  Includes self-reported complementary and integrative therapy use such as but not limited to massage, acupuncture, acupressure, chiropractic, mind-body therapies (e.g. Reiki), guided imagery, and others.
Adverse Events | 2, 4, 6, months
  Participant self-report of any new or worsening health issue while participating in the study. Participants will also be asked to report potential side effects by choosing from a list of known potential risks of exercise and mindfulness interventions.
Sleep Disturbance | Baseline, 2, 6 months
  Sleep disturbance will be measured using the PROMIS 6-item short form v1.0 which measures sleep quality on a 1 to 5 scale from very poor to very good in addition to agreement with statements on sleep quality on a 1 to 5 scale.
Sleep Duration | Baseline, 2, 6 months
  Participant's will self-report their average amount of sleep per night in the past month in hours and minutes.
Anxiety | Baseline, 2, 6 months
  Anxiety will be measured using the Generalized Anxiety Disorder-2 survey (GAD-2) which includes 2 questions that are summed for a total score that can range from 0 to 6.
Depression | Baseline, 2, 6 months
  Depression will be measured using the Patient Health Questionnaire-2 (PHQ-2) which includes 2 questions that are summed for a total score that can range from 0 to 6.
Participation in Social Roles and Activities | Baseline, 2, 6 months
  Measured using the PROMIS 4-item short form v2.0 which measures frequency of trouble doing activities for leisure, work, or with family or friends on a 1 to 5 scale.
Substance Use | Baseline, 2, 6 months
  Measured using the Tobacco, Alcohol, Prescription medications, and other Substance (TAPS) survey. The TAPS is comprised of a 4-item screen for substance use.

CONTACTS AND LOCATIONS:
Overall Officials: Roni L Evans, DC, MS, PhD, Principal Investigator — University of Minnesota; Brent Leininger, DC, MS, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
The study data will be submitted to a generalist repository that is participating in the NIH Generalist Repository Ecosystem Initiative. Demographic and clinical outcome measures will be collected and shared using common data elements (CDEs ) from the NIH / HEAL CDE repository. Variable naming and permissible response values will be harmonized according to CDEs data dictionary specifications. Documentation to be made publicly available to the research community and will include: 1. The study protocol; 2. informed consent form; 3. data collection forms/case report forms; 4. data dictionary.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Scientific data included in published manuscripts will be available at the time of publication; all other generated scientific data will be shared no later than the end of the award. The study data will be stored in the repository for at least 5 years.
Access Criteria: Data will be shared as allowed by the informed consents and institutional certification. Controlled Access will follow Data Use Limitations (DULs) to maximize the appropriate sharing of scientific data and protect research participants' privacy and confidentiality. Data will only be made available to the requester by the data repository after approval of the request by the data repository's independent review panel process.

REFERENCES:
- See also: Related Info — https://www.partners4pain.org